CLINICAL TRIAL: NCT00245193
Title: Motivationally-Enhanced Brief Interpersonal Psychotherapy for Depressed Mothers of Ill Children (MI-IPT-B-II)
Brief Title: Motivationally-Enhanced Brief Interpersonal Psychotherapy for Depressed Mothers of Ill Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23MH064518 (NIH); DSIR 8K-RTAT
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Depression
Keywords: Major Depression
MeSH Terms: conditions — Depression; Depressive Disorder, Major

INTERVENTIONS:
Behavioral: Motivationally-Enhanced Interpersonal Psychotherapy

SUMMARY:
This study will investigate the effectiveness of motivationally-enhanced brief interpersonal psychotherapy (MI-IPT-B) in treating depression in mothers who bring their children to a child mental health clinic for psychiatric treatment.

DETAILED DESCRIPTION:
Depression is a serious illness and is common in mothers who have children facing an illness. Research has shown that these mothers, in particular, need better coping skills and ways to relieve depressive symptoms. Helping mothers of ill children achieve better mental health may also be beneficial to their children. Studies have shown that psychotherapy is an effective treatment for depression, and often results in long-term improvements in depressive symptoms. This study will investigate the effectiveness of MI-IPT-B in treating depression in mothers who bring their children to a child mental health clinic for psychiatric treatment.

Participants in this open label study will be randomly assigned to receive either MI-IPT-B or facilitated referral to treatment as usual (F-TAU). Participants in both groups will undergo the same screening procedures following assignment to an intervention. The MI-IPT-B group will also receive one session of motivational therapy at the time of the initial screening procedures. Participants assigned to receive MI-IPT-B will report to the study site once weekly for therapy. This type of therapy will focus on improving the participants' relationships with their peers and the way that they perceive themselves. The F-TAU group will receive a referral for standard mental health care within the community health system. Both treatments will last 8 weeks. All participants will return to the study site at Week 14 and Month 6 for follow-up assessments of depressive symptoms.

ELIGIBILITY:
Inclusion Criteria

* Biological or adoptive mother whose child between the ages of 6 and 18 is treated in the Services for Teens at Risk (STAR) Center or the Center for Children and Families (CCF)
* Mother lives with and has custody of the child receiving treatment
* Meets DSM-IV criteria for current unipolar depressive disorder (e.g., dysthymic disorder, depressive disorder, or single or recurrent episodes of major depressive disorder)
* Score of greater than 16 on the Beck Depression Inventory
* Score of greater than 15 on the Hamilton Rating Scale for Depression (17-item)
* Willingness to maintain existing stable dose of antidepressant medication throughout the study if currently on medication and still experiencing symptoms of depression
* Willingness of child (treated in STAR clinic or CCF) to give informed consent

Exclusion Criteria:

* Currently receiving antidepressant medication at sub-therapeutic doses or at therapeutic doses but for an inadequate period of time to assess response
* Current dose of medication has not been stable for at least 8 weeks prior to study enrollment
* Suicidal or homicidal
* Requires hospitalization
* At risk for child abuse or neglect and requires intervention
* Simultaneous psychotic disorder or organic mental disorder
* History of drug or alcohol abuse within 6 months of study enrollment
* History of a prior manic episode
* Significant medical illness that might explain depressive symptoms (e.g., epilepsy, autoimmune disorders, liver dysfunction, unstable endocrine disease)
* Not fluent in English
* Severe cognitive deficits that would interfere with psychotherapy treatment
* Currently receiving another form of individual psychotherapy or couples therapy (except for participation in a support group, such as Alcoholics Anonymous)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-04; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Score on the Hamilton Rating Scale for Depression; measured at baseline, Week 14, and Month 6

SECONDARY OUTCOMES:
Score on the Beck Depression Inventory; measured at baseline, Week 14, and Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Holly Swartz, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States